CLINICAL TRIAL: NCT00483431
Title: Dose-finding Study for Vitamin K2 in Human Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEC 07-3-014
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2009-03

CONDITIONS: Vitamin K-status
Keywords: vitamin K2; dosis-response; osteocalcin; matrix-gla protein
MeSH Terms: interventions — menaquinone 7

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- PLACEBO (Placebo Comparator): MK7 dosage 0 mcg, 4 capsules, orally, daily for 12 weeks.
  Interventions: Dietary Supplement: Placebo
- MK7_10 (Active Comparator): MK7 dosage 10 mcg, 1 capsule of 10 mcg and 3 placebo-capsules, orally, daily for 12 weeks.
  Interventions: Dietary Supplement: MK7
- MK7_20 (Active Comparator): MK7 dosage 20 mcg, 2 capsules of 10 mcg and 2 placebo-capsules, orally, daily for 12 weeks.
  Interventions: Dietary Supplement: MK7
- MK7_45 (Active Comparator): MK7 dosage 45 mcg, 1 capsules of 45 mcg and 3 placebo-capsules, orally, daily for 12 weeks.
  Interventions: Dietary Supplement: MK7
- MK7_90 (Active Comparator): MK7 dosage 90 mcg, 2 capsules of 45 mcg and 2 placebo-capsules, orally, daily for 12 weeks.
  Interventions: Dietary Supplement: MK7
- MK7_180 (Active Comparator): MK7 dosage 180 mcg, 4 capsules of 45 mcg, orally, daily for 12 weeks.
  Interventions: Dietary Supplement: MK7
- MK7_360 (Active Comparator): MK7 dosage 360 mcg, 1 capsule of 360 mcg and 3 placebo-capsules, orally, daily for 12 weeks.
  Interventions: Dietary Supplement: MK7

INTERVENTIONS:
Dietary Supplement: Placebo
  Arms: PLACEBO
Dietary Supplement: MK7
  Other Names: Menaquinone-7
  Arms: MK7_10; MK7_180; MK7_20; MK7_360; MK7_45; MK7_90

SUMMARY:
Earlier studies have shown that high vitamin K-intake leads to improved bone and vascular health by increased carboxylation of Gla-proteins in these tissues. From all K-vitamins, Menaquinone-7 (MK7) has been identified as the most effective cofactor for the carboxylation reaction of Gla-proteins such as osteocalcin and matrix-gla protein. The question remains which dosage of MK7 leads to optimal carboxylation levels of these proteins.

The primary objective of this double-blind randomized intervention study is to establish the optimal dose of MK7 for carboxylation of the vitamin K-dependent proteins osteocalcin in bone and matrix-gla protein in the vessel wall. The optimal dose will be the concentration at which osteocalcin and matrix-gla protein are > 90% in the active (=carboxylated) form.

DETAILED DESCRIPTION:
This study is a double-blind randomized intervention study. In total 42 healthy volunteers (men and women) between 18 and 45 years will be recruited among the Maastricht University community (coworkers/students) and randomized into one of the following groups:

Placebo, 10 mcg MK7, 20 mcg MK7, 45 mcg MK7, 90 mcg MK7, 180 mcg MK7, 360 mcg MK7.

Each group will consist of 6 volunteers with approximately equal numbers of men and women (3 men / 3 women). A double-blind design of the study is chosen to avoid the occurrence of bias during the study. The randomization procedure will be performed by an investigator who is not involved in the coordination of the study and will generate specific randomization codes for each subject. After randomization, the volunteers consume the indicated amount of capsules once daily with either breakfast of dinner during a period of 12 weeks.

During the first week, blood samples of the volunteers will be collected at day 0, 1, 3 and 7 to study immediate effects on carboxylation of OC and MGP. After the first week, blood samples will be drawn every first day of week 2, 4, 6, 8, 10, and 12.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female adults between 18 and 45 years of age.
* Subjects of normal body weight and height according to BMI < 30
* Subject has given written consent to take part in the study

Exclusion Criteria:

* Subjects with (a history of) metabolic or gastrointestinal disease
* Subject with (a history of) soy allergy
* Subjects using vitamin supplements containing vitamin K
* Subjects presenting chronic inflammatory diseases
* Subjects receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters
* Subjects receiving corticoϊd treatment
* Subjects using oral anticoagulants

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2007-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
undercarboxylated osteocalcin (ucOC) | 12 weeks
  UcOC will be assessed by making use of a sandwich ELISA (in ng/ml)

SECONDARY OUTCOMES:
carboxylated osteocalcin (cOC) | 12 weeks
  cOC will be assessed by making use of a sandwich ELISA (in ng/ml)
undercarboxylated matrix-gla protein (ucMGP) | 12 weeks
  ucMGP will be assessed by making use of a sandwich ELISA (in pM)

CONTACTS AND LOCATIONS:
Overall Officials: Cees Vermeer, PhD, Principal Investigator — Maastricht University
Locations (1):
- VitaK BV / University of Maastricht, Maastricht, PO Box 616, Netherlands

REFERENCES:
- [Derived] Theuwissen E, Cranenburg EC, Knapen MH, Magdeleyns EJ, Teunissen KJ, Schurgers LJ, Smit E, Vermeer C. Low-dose menaquinone-7 supplementation improved extra-hepatic vitamin K status, but had no effect on thrombin generation in healthy subjects. Br J Nutr. 2012 Nov 14;108(9):1652-7. doi: 10.1017/S0007114511007185. Epub 2012 Jan 31. PMID 22289649
- [Derived] Knapen MH, Schurgers LJ, Shearer MJ, Newman P, Theuwissen E, Vermeer C. Association of vitamin K status with adiponectin and body composition in healthy subjects: uncarboxylated osteocalcin is not associated with fat mass and body weight. Br J Nutr. 2012 Sep 28;108(6):1017-24. doi: 10.1017/S000711451100626X. Epub 2011 Dec 5. PMID 22136751